CLINICAL TRIAL: NCT05686369
Title: A Decentralized Home-Based Study To Investigate Novel Objective Biomarker Of Gluten-Mediated Symptoms Using A Wearable Biosensor And A Mobile Platform In Celiac Disease Participants With And Without Gluten Challenge (CeDar ROSE Study)
Brief Title: A Decentralized Home-Based Study To Investigate Novel Objective Biomarker Of Gluten-Mediated Symptoms In Celiac Disease Participants (CeDar ROSE Study)
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: DQB002UZ
Record Dates: First submitted 2022-11-08; First posted 2023-01-17 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Well-controlled Celiac Disease: Cohort A: Well-controlled celiac disease participants who should be asymptomatic or mildly symptomatic
- Cohort B: Non-Responsive Celiac Disease: Cohort B: Celiac disease participants with persistent symptoms who are known to be symptomatic and show positivity to serum auto-antibodies even though participants have been adhering to gluten-free diet

SUMMARY:
This is a decentralized study to primarily explore a novel objective digital biomarker (i.e., Gluten Dependency Index) for celiac disease-related responses triggered by gluten exposure using a wearable biosensor. This study also explores a novel objective blood biomarker specific to celiac disease activity and evaluates participant symptoms, lifestyle and an objective comprehensive measurement (e.g., activity, stress and sleep) in celiac disease participants.

Approximately 170 well-controlled celiac disease participants (Cohort A) and 40 celiac disease participants with persistent symptoms (Cohort B) will be monitored for 13 and 8 weeks in the observation period, respectively, in a home-based setting using the wearable biosensor along with a mobile platform including some electronic questionnaires.

The wearable biosensor continuously records biosensor data. These data will be used to develop a new algorithm for Gluten Dependency Index and calculate the Gluten Dependency Index, Activity Value, Stress Value, or Sleep Time. Participants will report celiac disease-related symptoms, diet (including any accidental gluten exposures), exercise, menstruation questionnaires in CDSD and mobile platform questionnaire (MPFQ), which is originally designed by the Sponsor.

All participants both in Cohort A and B are required to maintain gluten-free diet throughout the study. Only participant who are enrolled in Cohort A will be required gluten challenge.

ELIGIBILITY:
Inclusion Criteria:

[Cohort A and B]

* History of medically diagnosed celiac disease based on biopsies and positive celiac serology.
* Be on a GFD for at least 12 months
* Willing and able to adhere to use and management of the wearable device
* Willingness to comply with home-based approach and visits by a HN professional [Cohort A only]
* Experienced at most mild symptoms of celiac disease
* Willingness to consume food containing up to 6 g of gluten protein per challenge day and up to 18 g of gluten protein in total during the study [Cohort B only]
* Experienced at least 2 different gluten-related symptoms (e.g., diarrhea, abdominal pain, bloating, nausea, tiredness) or 1 gluten-related symptom occurred twice within the month before screening, and at screening were required to have a qualifying score as moderate or severe on at least one symptom on the CDSD in the 14 days recording period.
* Positive for any of the 3 serology tests, tissue - transglutaminase-2-IgA [tTG2-IgA] (≥4 U/mL), deamidated gliadin peptide-IgA [DGP-IgA] (≥20 U/mL), or deamidated gliadin peptide-IgG [DGP-IgG] (≥20U/mL)

Exclusion Criteria:

[Cohort A and B] Refractory celiac disease [Cohort A] Positive for any of the 3 serology tests

* Tissue transglutaminase-2 [tTG2-IgA] (≥10 U/mL; normal range: 0-3.99 U/mL) prior to the observation period, but weak positive (4-10 U/mL) can be enrolled in this study.
* Deamidated gliadin peptide-IgA [DGP-IgA], and deamidated gliadin peptide-IgG [DGP-IgG] prior to the observation period, but weak positive (20-30 U/mL) can be enrolled.

History of IgE-mediated reactions to wheat, barley, rye, or other ingredients in the gluten products used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A: Well-controlled celiac disease participants who should be asymptomatic or mildly symptomatic Cohort B: Celiac disease participants with persistent symptoms who are known to be symptomatic and show positivity to serum auto-antibodies even though participants have been adhering to gluten-free diet
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
The concordance between the novel digital biomarker and the presence of celiac disease-related symptoms | up to 13 weeks

SECONDARY OUTCOMES:
Correlations between the comprehensive measurement and the scores of patient reported outcomes | up to 13 weeks
  Correlations between the comprehensive measurement and the scores of Celiac Disease Symptom Diary (CDSD), 36-Item Short Form Survey (SF-36), or Celiac Disease-related Quality of Life (CDQOL)
The comprehensive measurement | up to 13 weeks
  The comprehensive measurement objectively evaluated by wearable biosensor
The scores of Celiac Disease Symptom Diary (CDSD) | up to 13 weeks
  Scoring rate for celiac disease symptoms Minimum: Non Maximum: Very severe
The scores of Short Form 36 (SF-36) | up to 13 weeks
  Scoring rate for quality of life (higher score-better quality of life) Minimum: 0 Maximum: 100
The scores of Celiac Disease-related Quality of Life (CDQOL) | up to 13 weeks
  Scoring rate for quality of life in celiac disease participants Minimum: 1 (total disagreement) Maximum: 5 (total agreement)
Adverse events | up to 13 weeks
  Incidence and severity of adverse events
Adverse events' relationship to gluten exposure | up to 13 weeks
  Incidence and severity of adverse events' relationship to gluten exposure
Safety as assessed by systolic and diastolic by blood pressure | up to 13 weeks
  Abnormality in blood pressure
Safety as assessed by body temperature | up to 13 weeks
  Abnormality in body temperature
Safety as assessed by pulse rate | up to 13 weeks
  Abnormality in pulse rate
Safety as assessed by respiratory rate | up to 13 weeks
  Abnormality in respiratory rate
Safety as assessed by percutaneous oxygen saturation | up to 13 weeks
  Abnormality in percutaneous oxygen saturation
Safety as assessed by hematology test with counting blood cells | up to 13 weeks
  Incidence of hematology abnormalities
Safety as assessed by blood chemistry test with measuring chemicals | up to 13 weeks
  Incidence of blood chemistry abnormalities
Safety as assessed by coagulation testing with thrombolytic capacity measurement | up to 13 weeks
  Incidence of coagulation abnormalities
Safety as assessed by urinalysis test with examining the visual, chemical and microscopic aspects | up to 13 weeks
  Incidence of urinalysis abnormalities
Safety as assessed by Electrocardiograms (QT interval) | up to 13 weeks
  Abnormality in QT interval
Safety as assessed by Electrocardiograms (heart rate) | up to 13 weeks
  Abnormality in heart rate
Celiac disease serology levels | up to 13 weeks
  Serology levels about tissue transglutaminase-2-IgA (tTG2-IgA; unit/mL)
Celiac disease serology levels | up to 13 weeks
  Serology levels about Deamidated gliadin peptide-IgA (DGP-IgA; unit), and deamidated gliadin peptide-IgG (DGP-IgG; unit)
3072 Blood biomarkers profile | up to 13 weeks
  3072 Blood biomarkers profile measured by proteomics in well-controlled celiac disease participants (Cohort A) and in celiac disease participants with persistent symptoms (Cohort B)
48 Blood biomarker profile | up to 13 weeks
  48 Blood biomarkers profile measured by proteomics in well-controlled celiac disease participants (Cohort A) and in celiac disease participants with persistent symptoms (Cohort B)
Change from baseline in 3072 blood biomarkers profile (Cohort A only) | up to 13 weeks
  Change from baseline in 3072 blood biomarker profile measured by proteomics after gluten/sham gluten challenge (Cohort A only)
Change from baseline in 48 blood biomarkers profile (Cohort A only) | up to 13 weeks
  Change from baseline in 48 blood biomarkers profile measured by proteomics after gluten/sham gluten challenge (Cohort A only)
The incidence of novel digital biomarker (Cohort B only) | up to 13 weeks
  The incidence of novel digital biomarker established in Cohort A (Cohort B only)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (1):
- Science 37, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).